CLINICAL TRIAL: NCT04353557
Title: Monitoring Circulating Tumor DNA in Patients With Early Stage Breast Cancer
Brief Title: ctDNA Monitoring in Early Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Geneplus-Beijing Co. Ltd. (Industry)
Collaborators: Army Medical University, China (Other)
Responsible Party: Sponsor
Other Study IDs: Geneplus2020BC01
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
Keywords: ctDNA
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor and plasma specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a observational, single center study, monitoring the circulating tumor DNA (ctDNA) in patients with early breast cancer and assessing the prognostic value and treatment outcome monitoring of ctDNA.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 80 years old
2. Histologically proven primary breast cancer with clinical stage I-III
3. Patients with neoadjuvant therapy, and/or radical surgery/breast conserving surgery, adjuvant chemotherapy and target therapy (Her2+), radiotherapy (if indicated).
4. Expected to achieve R0 resection.
5. Estimated lifetime is more than 3 months.
6. Signed Informed Consent Form
7. Consent to provide research blood samples.

Exclusion Criteria:

1. Patients intended to receive adjuvant chemotherapy with Eastern Cooperative Oncology Group (ECOG) performance status 3, 4 or 5.
2. Patients intended to receive postoperative radiotherapy with Eastern Cooperative Oncology Group (ECOG) performance status 5.
3. Prior diagnosis of cancer in the previous 5 years, other than for basal cell carcinoma of the skin or cervical carcinoma in situ.
4. Presence of any systemic illness incompatible with participation in the clinical trial or inability to provide written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage I-III breast cancer who planed to receive curative-intent treatment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-11-29 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Positive ctDNA detection at first post-operative timepoint | 1 month post-surgery
  The proportion of patients with ctDNA positivity as assessed by the blood sample taken at first post-operative timepoint

SECONDARY OUTCOMES:
Positive ctDNA detection at post-operative timepoints | 6/12/18/24/30 months
  The proportion of patients with ctDNA positivity as assessed by the blood sample taken at other post-operative timepoints
Association between ctDNA detection and time to recurrence | 1 month post-surgery
  Time to recurrence of subgroups with detectable ctDNA and undetectable ctDNA comparison.
Association between ctDNA detection and time to recurrence | 6/12/18/24/30 months
  Time to recurrence of subgroups with detectable ctDNA and undetectable ctDNA

CONTACTS AND LOCATIONS:
Locations (1):
- Army Medical Center of PLA, China, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No